CLINICAL TRIAL: NCT06150781
Title: GENESIS: AIMOVIG® Pregnancy Exposure Registry
Brief Title: Aimovig Pregnancy Exposure Registry
Status: Recruiting | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20180125
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Erenumab-Aooe; AIMOVIG®
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Erenumab-aooe-exposed: Pregnant women with confirmed migraine who received erenumab-aooe before or during pregnancy will qualify to be included in the cohort. Dosing and treatment duration of erenumab-aooe as part of this observational study is at the discretion of the healthcare provider (HCP) in accordance with local clinical practice and local labeling.
  Interventions: Drug: erenumab-aooe
- Erenumab-aooe-unexposed (Internal Comparator): Pregnant women with clinically confirmed migraine who were not exposed to erenumab-aooe before or during pregnancy will be included in the internal comparator cohort.
- Women Without Migraine (External Comparator): Pregnant woman without migraine will be included in this cohort as external comparator. The Metropolitan Atlanta Congenital Defects Program (MACDP) birth defects classification system will be used to characterize major and minor congenital malformations for this study.

INTERVENTIONS:
Drug: erenumab-aooe — Dose and treatment duration will be advised by the HCP
  Other Names: Aimovig®
  Groups: Erenumab-aooe-exposed

SUMMARY:
The primary objective of this study is to estimate the proportion of major congenital malformations in infants of women with migraine exposed to erenumab-aooe during pregnancy compared to infants of women with migraine unexposed to erenumeb-aooe.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older (at time of signing the informed consent)
* Currently pregnant
* The outcome of the pregnancy must not be known
* Confirmed clinical diagnosis of migraine

Exclusion Criteria:

* Women currently participating in another investigational device or investigational drug study, currently taking an investigational medicinal product, or having taken an investigational product within 3 months prior to last menstrual period (LMP) or during pregnancy. Other investigational procedures while participating in this study are excluded.
* Women exposed to any medications that target the calcitonin gene-related peptide (CGRP) pathway (ie, CGRP monoclonal antibody [mAb] or gepants) in the period from 5 half-lives prior to LMP through the end of pregnancy.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 2842 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Number of Infants Experiencing Major Congenital Malformations | Up to 52 Weeks

SECONDARY OUTCOMES:
Number of Women with Pregnancy Complications Following Erenumab-aooe Administration | Week 52
Number of Women Experiencing Spontaneous Abortion, Still Birth, Elective Termination, and Preterm Birth | Up to Approximately 38 Weeks
Percentage of Infants of Women Exposed to Erenumab-aooe who are Small-for-gestational age | Up to Approximately 38 Weeks
Percentage of Infants of Women Exposed to Erenumab-aooe Experiencing Minor Congenital Malformations | Up to Week 52
Percentage of Infants of Women Exposed to Erenumab-aooe with Postnatal Growth and Development Deficiency Through the First Year of life | Up to Week 52
Percentage of Participants with Maternal Outcomes | Up to Approximately 38 Weeks
  Pregnancy outcomes: elective or spontaneous termination, fetal death, preterm birth.
Percentage of Participants with Fetal Outcomes | Up to Approximately 38 Weeks
  Pregnancy outcomes: elective or spontaneous termination, fetal death, preterm birth.
Percentage of Participants with Infant Outcomes | Up to Week 52
  Infant outcomes: minor congenital malformations, size for gestational age, low birth weight, postnatal growth and development.
Frequency of Major Congenital Malformations of Women with Migraine Exposed to Erenumab-aooe During Pregnancy with Women Representing the Prevalence of Birth Defects in the General Population (External Comparator) | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- IQVIA Virtual Site, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com